CLINICAL TRIAL: NCT04724018
Title: Combinations of Sacituzumab Govitecan Plus Enfortumab Vedotin and Pembrolizumab for Metastatic Urothelial Carcinoma: the Double Antibody Drug Conjugate (DAD) and Double Antibody Drug Conjugate With Immunotherapy (DAD-IO) Phase I/II Trial
Brief Title: Sacituzumab Govitecan Plus EV in Metastatic UC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Bradley A. McGregor, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-614
Record Dates: First submitted 2021-01-20; First posted 2021-01-26 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Urothelial Cancer; Metastatic Urothelial Carcinoma; Metastatic Urothelial Carcinoma of the Renal Pelvis and Ureter; Bladder Cancer
Keywords: Urothelial cancer; Metastatic Urothelial Carcinoma; Metastatic Urothelial Carcinoma of the Renal Pelvis and Ureter; Bladder Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — sacituzumab govitecan; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation Sacituzumab Govitecan (SG) and Enfortumab vedotin-ejfv (EV) (Experimental): Participants will be given the study drugs Enfortumab Vedotin and then Sacituzumab Govitecan on Days 1 and 8 of a 21-day study cycle. Dose escalation and de-escalation for the Sacituzumab Govitecan (SG) and Enfortumab vedotin-ejfv (EV) combination will be guided using the Bayesian optimal interval (BOIN) design with up to 4 dose level escalations.
  Interventions: Drug: Sacituzumab Govitecan (SG); Drug: Enfortumab vedotin-ejfv (EV)
- Dose Expansion Sacituzumab Govitecan (SG) and Enfortumab vedotin-ejfv (EV) (Experimental): Participants will be given the study drugs Enfortumab Vedotin and then Sacituzumab Govitecan on Days 1 and 8 of each 21-day study cycle. Three dose levels of this drug combination will be studied with 3-18 patients per dose level depending on treatment-related dose limiting toxicities.
  Interventions: Drug: Sacituzumab Govitecan (SG); Drug: Enfortumab vedotin-ejfv (EV)
- Sacituzumab Govitecan (SG) and Enfortumab vedotin-ejfv (EV) and Pembrolizumab (Experimental): Participants will be given a triplet regimen of Enfortumab Vedotin 1.25mg/kg, Sacituzumab Govitecan 7.5mg/kg (D1 and D8 every three weeks), and Pembrolizumab 200mg (D1 every 3 weeks) or 400 mg (D1 every 6 weeks) as a front-line therapy. Dose reductions of Enfortumab Vedotin to 1, 0.75 and 0.5 mg/kg will be permitted while Sacituzumab Govitecan can be dose reduced to 5 mg/kg. No dose reductions of Pembrolizumab are permitted. Following C1D1, drugs may be held independently per investigator discretion. A safety run-in will be conducted for the first 12 patients to evaluate the tolerability of the triplet regimen using Bayesian toxicity monitoring (BTOX). The first stage will enroll 6 patients, and if there are 2 or fewer DLTs, then next 6 patients will be enrolled. The study will be halted if there are 5 or more DLTs observed among the total of 12 evaluable patients.
  Interventions: Drug: Sacituzumab Govitecan (SG); Drug: Enfortumab vedotin-ejfv (EV); Drug: Pembrolizumab

INTERVENTIONS:
Drug: Sacituzumab Govitecan (SG) — Intravenous infusion
  Other Names: Trodelvy
Drug: Enfortumab vedotin-ejfv (EV) — Intravenous infusion
  Other Names: Padcev
Drug: Pembrolizumab — Intravenous infusion
  Other Names: Keytruda
  Arms: Sacituzumab Govitecan (SG) and Enfortumab vedotin-ejfv (EV) and Pembrolizumab

SUMMARY:
Phase I of this research study will assess what doses of Sacituzumab Govitecan and Enfortumab Vedotin can be safely combined in the treatment of metastatic urothelial carcinoma (mUC). In Phase II of the study, patients in one of the two cohorts will receive Sacituzumab Govitecan, Enfortumab Vedotin, and Pembrolizumab to assess the efficacy of this drug combination.

The names of the study drugs in these investigational combinations are:

* Enfortumab Vedotin
* Sacituzumab Govitecan
* Pembrolizumab

DETAILED DESCRIPTION:
Phase I of this study was a single-center, open-label, nonrandomized phase I trial testing the safety and efficacy as well as defining the appropriate dose for future studies of Sacituzumab Govitecan and Enfortumab for people with metastatic urothelial carcinoma (mUC) progressing on platinum-based chemotherapy and PD1/L1 inhibitors.

The U.S. Food and Drug Administration (FDA) has approved Enfortumab Vedotin for the treatment of metastatic urothelial carcinoma (mUC) (bladder cancer). The FDA has not approved Sacituzumab Govitecan for metastatic urothelial carcinoma (mUC) (bladder cancer) but it has been approved for other uses. The FDA has approved Sacituzumab Govitecan to treat a type of breast cancer at this time. Sacituzumab Govitecan has appeared promising in patients with bladder cancer that has spread and works by a different mechanism than Enfortumab Vedotin. Therefore, the researchers believe that combining these 2 drugs may control the cancer better than each drug does on its own.

This will be done through testing different combinations and checking for serious side effects; if there are no serious side effects a different dose combination will be explored. Once the best combination has been determined, the study will expand to a phase 2 trial looking how effective (how well the drug works)the combination in slowing down the growth of metastatic urothelial carcinoma (mUC) progressing on platinum-based chemotherapy and PD1/L1 inhibitors and in combination with PD1/PDL1 inhibitors in treatment naive disease.

Phase II of this study is a multicenter phase 2 trial to to test the efficacy of Sacituzumab Govitecan in combination with Enfortumab Vedotin in patients with treatment refractory urothelial carcinoma (Cohort A). Phase II will also study the efficacy of the combination of Enfortumab Vedotin, Sacituzumab Govitecan, and Pembrolizumab in patients who have not yet received systemic therapy for metastatic carcinoma and are more than 6 months from completion of any immunotherapy in the perioperative setting (Cohort B).

The research study procedures include screening for eligibility, study treatment, and safety follow-up visits, in addition to general health status follow-up after study treatment.

Participants will receive study treatment for as long as they do not have serious side effects and their disease does not get worse. However, the duration may vary depending on how long the treatment works to control the cancer and how someone's body tolerates the side effects.

Gilea, a pharmaceutical company, is supporting this research study by providing funding for the research study, tests required for research purposes only, and the study drug Sacituzumab Govitecan.

It is expected that up to 24 people will take part in Phase I of this research study and up to 41 people will take part in each of the two Phase II cohorts.

ELIGIBILITY:
Phase II Study Cohort A (dose expansion study to assess efficacy of Sacituzumab Govitecan (SG) and Enfortumab vedotin-ejfv (EV) combination)

Inclusion Criteria:

* Participants must have histologically documented confirmed predominant urothelial carcinoma (i.e. of the bladder, renal pelvis, ureter or urethra). Patients with squamous differentiation or mixed cell types are eligible if the urothelial component is more than 50%; small-cell carcinoma is not allowed. Patients with locally advanced unresectable disease are eligible.
* Patient who are cisplatin eligible must have received prior treatment with platinum containing therapy defined as within the adjuvant/neoadjuvant setting with ≥ ypT2 disease at surgery or recurrent or progressive disease within 12 months or receiving treatment with platinum in locally advanced or metastatic setting. In addition, they must have received a checkpoint inhibitor (CPI) in locally advanced or metastatic urothelial cancer setting. Patients who received CPI therapy in the neoadjuvant/adjuvant setting and had recurrent or progressive disease either during or within 12 months of therapy completion are eligible. A CPI is defined as a PD-1 or PD-L1 inhibitor.
* Patients who are cisplatin-ineligible need only have progressed on or since one line of therapy defined as therapy given in the adjuvant/neoadjuvant setting within 12 months of progression or receiving therapy for locally advanced or metastatic disease
* Patient must be progressing on or since most recent therapy
* Age ≥18 years. Children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG performance status 0-1.
* Participants must have adequate organ and marrow function as defined below:
* Leukocytes ≥3,000/mcL
* Absolute neutrophil count ≥1,500/mcL
* Platelets ≥100,000/mcL
* Total bilirubin ≤ institutional upper limit of normal (ULN)
* AST(SGOT)/ALT(SGPT) ≤2.5x institutional ULN OR
* ≤5x ULN with liver metastases and serum albumin > 3 g/dL
* Glomerular filtration rate (GFR) ≥30 mL/min/1.73 m2 (by Cockcroft Gault formula)
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Have measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) as per response evaluation criteria in solid tumors version 1.1 (RECIST 1.1 criteria). Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 6 months after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >2 years
* The effects of SG and EV on the developing human fetus are unknown. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and 6 months after last study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study and up to 6 months after last study drug dose, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of SG administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria at Screening/Day 1 of treatment will not be enrolled in the study.

* Women who are pregnant or lactating. Pregnant women are excluded from this study because SG and EV have potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with EV or SG, breastfeeding should be discontinued if the mother is treated on protocol.
* Have had a prior anti-cancer biologic agent (including immune checkpoint inhibitors) within 4 weeks prior to Cycle 1 Day 1 (C1D1) or have had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to C1D1. Subjects participating in observational studies are eligible.
* Presence of any toxicities attributed to prior anti-cancer therapy that are not resolved to Grade 1 or baseline that could impose serious risk for complications before administration of study drug agent
* Note: If subjects received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Have previously received topoisomerase 1 inhibitors, SG or EV
* Have an active second malignancy. Subjects with a history of malignancy that have been completely treated, with no evidence of active cancer for 3 years prior to start of therapy on trial (Cycle 1 Day 1 [C1D1]), or subjects with surgically-cured tumors with low risk of recurrence are allowed to enroll.
* Have known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they have stable CNS disease for at least 4 weeks prior to the first dose of study drug and all neurologic symptoms have returned to baseline, have no evidence of new or enlarging brain metastases, and are taking ≤20 mg/day of prednisone or its equivalent. All subjects with carcinomatous meningitis are excluded regardless of clinical stability.
* Have active cardiac disease, defined as:
* Myocardial infarction or unstable angina pectoris within 6 months prior to C1D1
* History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation
* New York Heart Association (NYHA) Class III or greater congestive heart failure or left ventricular ejection fraction of < 40%
* Have active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or gastrointestinal (GI) perforation within 6 months of C1D1
* Have active serious infection requiring antibiotics (Contact sponsor-investigator for clarification)
* Have other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
* Patients with conditions requiring high doses of steroids (>10 mg/day of prednisone or equivalent) or other immunosuppressive medications are excluded. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.
* History of idiopathic pulmonary fibrosis; organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Participants who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to EV or SG or any excipient contained in the drug formulations (including 2 (N morpholino) ethane sulfonic acid (MES), histidine, treahalose dihydrate polysorbate 80 and polysorbate 20).
* Participants with uncontrolled intercurrent illness.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with uncontrolled diabetes. Uncontrolled diabetes is defined as hemoglobin A1C >8% or 7-8% with associated diabetes symptoms that are otherwise not explained
* Uncontrolled tumor related bone pain or impending spinal cord compression.

Phase II Study Cohort B (assessing Sacituzumab Govitecan (SG) + Enfortumab vedotin-ejfv (EV) + Pembrolizumab combination)

Inclusion Criteria:

* Participants must have histologically documented confirmed predominant urothelial carcinoma (i.e. of the bladder, renal pelvis, ureter or urethra). Patients with squamous differentiation or mixed cell types are eligible if the transitional component is more than 50%; small-cell carcinoma is not allowed. Patients with locally advanced unresectable disease are eligible.
* No prior therapy for metastatic urothelial carcinoma. Therapy in the perioperative setting is allowed with no time restrictions on platinum dosing. Prior immunotherapy is allowed provided it has been > 6 months from last dose of immune checkpoint blockade.
* Age ≥18 years; children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG performance status 0-1.
* Participants must have adequate organ and marrow function as defined below:
* Leukocytes ≥3,000/mcL
* Absolute neutrophil count ≥1,500/mcL
* Platelets ≥100,000/mcL
* Total bilirubin ≤ institutional upper limit of normal (ULN)
* AST(SGOT)/ALT(SGPT) ≤2.5x institutional ULN OR
* ≤5x ULN with liver metastases and serum albumin > 3 g/dL
* Glomerular filtration rate (GFR) ≥30 mL/min/1.73 m2 (by Cockcroft Gault formula)
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Have measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) as per response evaluation criteria in solid tumors version 1.1 (RECIST 1.1 criteria). Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 6 months after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >2 years
* The effects of Pembrolizumab, SG and EV on the developing human fetus are unknown. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and 6 months after last study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study and up to 6 months after last study drug dose, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of SG administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria at Screening/Day 1 of treatment will not be enrolled in the study.

* Women who are pregnant or lactating. Pregnant women are excluded from this study because SG and EV have potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with EV or SG, breastfeeding should be discontinued if the mother is treated on protocol.
* Have had a prior anti-cancer biologic agent (including immune checkpoint inhibitors) or chemotherapy within 26 weeks prior to Cycle 1 Day 1 (C1D1) Subjects participating in observational studies are eligible.
* Have previously received topoisomerase 1 inhibitors, SG or EV
* Have an active second malignancy. Subjects with a history of malignancy that have been completely treated, with no evidence of active cancer for 3 years prior to start of therapy on trial (Cycle 1 Day 1 [C1D1]), or subjects with surgically-cured tumors with low risk of recurrence are allowed to enroll.
* Have known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they have stable CNS disease for at least 4 weeks prior to the first dose of study drug and all neurologic symptoms have returned to baseline, have no evidence of new or enlarging brain metastases, and are taking ≤10 mg/day of prednisone or its equivalent. All subjects with carcinomatous meningitis are excluded regardless of clinical stability.
* Have active cardiac disease, defined as:

  * Myocardial infarction or unstable angina pectoris within 6 months prior to C1D1
  * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation
* New York Heart Association (NYHA) Class III or greater congestive heart failure or left ventricular ejection fraction of < 40%
* Have active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or gastrointestinal (GI) perforation within 6 months of C1D1
* Have active serious infection requiring antibiotics (Contact sponsor PI or Co-PI for clarification)
* Have other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
* Patients with conditions requiring high doses of steroids (>10 mg/day of prednisone or equivalent) or other immunosuppressive medications are excluded. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.
* History idiopathic pulmonary fibrosis; organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Participants who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab, EV or SG or any excipient contained in the drug formulations (including 2 (N morpholino) ethane sulfonic acid (MES), histidine, treahalose dihydrate polysorbate 80 and polysorbate 20).
* Participants with uncontrolled intercurrent illness.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with uncontrolled diabetes. Uncontrolled diabetes is defined as hemoglobin A1C >8% or 7-8% with associated diabetes symptoms that are otherwise not explained
* Uncontrolled tumor related bone pain or impending spinal cord compression.
* History of autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).

  1. Replacement therapy (e.g., thyroxine, insulin, physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
  2. Brief (<7 days) use of systemic corticosteroids is allowed when use is considered standard of care.
  3. Subjects with vitiligo, psoriasis, type 1 diabetes mellitus, hypothyroidism, or resolved childhood asthma/atopy will not be excluded.
  4. Subjects requiring intermittent use of bronchodilators, inhaled steroids, or local steroid injections will not be excluded.
  5. Subjects with hypothyroidism that is stable with hormone replacement or Sjögren's syndrome will not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Sacituzumab Govitecan (SG) and Enfortumab vedotin-ejfv (EV) in Combination | 21 days
  The Maximum Tolerated Dose (MTD) in mg of Sacituzumab Govitecan (SG) and Enfortumab vedotin-ejfv (EV) in Combination is assessed.
Dose-limiting toxicity (DLT) of Sacituzumab Govitecan (SG) and Enfortumab Vedotin in combination | 21 days
  Treatment-Related Adverse Events are assessed by CTCAE v5.0 when administering Sacituzumab Govitecan (SG) and Enfortumab Vedotin (EV) in combination.
Efficacy of Sacituzumab Govitecan (SG) and Enfortumab Vedotin in combination | 21 days
  Study SG + EV combination to further refine the recommended dose and to assess the ORR (unconfirmed CR or PR) per RECIST Version 1.1 as determined by investigator for the combination of EV and SG in combination in patients with mUC progressing on platinum-based chemotherapy and PD1/L1 inhibitors.
Efficacy of Sacituzumab Govitecan (SG) and Enfortumab Vedotin and Pembrolizumab in combination | 21 days
  Study SG + EV + Pembrolizumab in combination to assess the ORR (unconfirmed CR or PR) per RECIST Version 1.1 as determined by investigator for the combination therapy of Pembrolizumab in combination with EV and SG in treatment-naïve patients with mUC.

SECONDARY OUTCOMES:
Sacituzumab Govitecan (SG) and Enfortumab Vedotin in combination objective response rate (ORR) | 21 days
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Sacituzumab Govitecan (SG) and Enfortumab Vedotin in combination rate of complete responses (CR) | 21 days
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Sacituzumab Govitecan (SG) and Enfortumab Vedotin in combination rate of partial responses (PR) | 21 days
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Sacituzumab Govitecan (SG) and Enfortumab Vedotin in combination rate of participants with progressive disease | 21 days
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Sacituzumab Govitecan (SG) and Enfortumab Vedotin in combination overall survival (OS) Rate | 21 days
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Sacituzumab Govitecan (SG) and Enfortumab Vedotin in combination expansion cohort progression-free survival. | 21 days
  Assessed as progression-free survival per investigator assessment.
Sacituzumab Govitecan (SG) and Enfortumab Vedotin in combination expansion cohort overall survival (OS) rate. | 21 days
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Sacituzumab Govitecan (SG) and Enfortumab Vedotin in combination expansion cohort safety assessment. | 21 days
  Treatment-Related Adverse Events are assessed by CTCAE v5.0 when administering Sacituzumab Govitecan (SG) and Enfortumab Vedotin (EV) in combination.
Sacituzumab Govitecan (SG) and Enfortumab Vedotin and Pembrolizumab in combination progression-free survival. | 21 days
  Assessed as progression-free survival per investigator assessment.
Sacituzumab Govitecan (SG) and Enfortumab Vedotin and Pembrolizumab in combination overall survival (OS) rate. | 21 days
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Sacituzumab Govitecan (SG) and Enfortumab Vedotin and Pembrolizumab in combination safety assessment. | 21 days
  Treatment-Related Adverse Events are assessed by CTCAE v5.0 when administering Sacituzumab Govitecan (SG) and Enfortumab Vedotin (EV) and Pembrolizumab in combination.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley A McGregor, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] McGregor BA, Sonpavde GP, Kwak L, Regan MM, Gao X, Hvidsten H, Mantia CM, Wei XX, Berchuck JE, Berg SA, Ravi PK, Michaelson MD, Choueiri TK, Bellmunt J. The Double Antibody Drug Conjugate (DAD) phase I trial: sacituzumab govitecan plus enfortumab vedotin for metastatic urothelial carcinoma. Ann Oncol. 2024 Jan;35(1):91-97. doi: 10.1016/j.annonc.2023.09.3114. Epub 2023 Oct 21. PMID 37871703